CLINICAL TRIAL: NCT03094455
Title: Action-Observation Therapy (AOT) and Information and Communications Technologies (ICT) for Home Rehabilitation of Hemiplegia
Brief Title: AOT and ICT for Hemiplegia
Acronym: Tele-UPCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: BioRobotics Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2011-02350053 AOT
Record Dates: First submitted 2017-03-16; First posted 2017-03-29 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Hemiplegia; Hemiplegic Cerebral Palsy
Keywords: Tele-rehabilitation; Action Observation; Mirror neurons; ICT
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: It will be a parallel RCT with a waitlist design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): AOT is based on the observation of meaningful actions followed by their execution
  Interventions: Other: Experimental group
- Control group (Other): Children will continue standard care for 3 weeks and then will receive the AOT as the Experimental group
  Interventions: Other: Experimental group

INTERVENTIONS:
Other: Experimental group — Observation of video sequences showing uni¬manual or bimanual goal-directed actions followed by the execution of the observed actions either with plegic upper limb for unimanual or with both upper limbs for bimanual actions.
  Other Names: AOT

SUMMARY:
A new rehabilitative approach, called AOT, based on the recent discovery of mirror neuron system (MNS), has been used with promising results on the Upper Limb (UL) function in some studies in children with Cerebral Palsy (CP).The purpose of the present trial is to provide evidence by a RCT that AOT is an effective rehabilitation tool in Children with Unilateral CP (UCP) and that its effects are greater than standard care. Assisting Hand Assessment is chosen as primary outcome measure and a sample size of 10 per group is required. The rehabilitation lasting 3 weeks will be provided at home by an ICT platform able to deliver, manage, monitor and measure a personalized AOT.

DETAILED DESCRIPTION:
A waitlist control, evaluator-blinded, randomized trial (RCT) will be conducted according to CONSORT guidelines. Each participant will be randomized to either:

1. Immediate intervention group (Experimental group). Children will receive immediately the system for 3 weeks.
2. Waitlist delayed intervention (Control group). Children will continue standard care for 3 weeks and then will receive the system as the Experimental group.

As such, all participants will receive the AOT training. The system will provide an in-home, individualized, intensive treatment based on the AOT. The system will be delivered at home and the children will perform a 60-minute training session 5 days a week for 3 consecutive weeks. For the Immediate intervention group, follow-up assessment (outcome measures) will be conducted before (T0) and post-intervention at 3 weeks (T1), and then 8 and 24 weeks after T1(T2 and T3). For the Waitlist group, the assessments will be conducted before T0 and 3 weeks after (T1) the standard care, then they will follow the same timeline of the first group (T1 plus, after the AOT intervention) and 8 and 24 weeks after T1 Puls (T2 and T3). The primary endpoint will be T1. Clinical assessments will be administered by a therapist blind to group assignment in each center. Scoring of videotaped clinical outcome measures will be performed by therapists blind to group allocation and assessment order.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of spastic UCP
* age between 15 and 20 years
* predominant spasticity at upper limb upper limb
* minimal ability to grasp and hold objects, also passively, with affected hand (House functional classification score 2 or more)
* sufficient cooperation, cognitive and communicative understanding to perform assessments and participate in the intervention
* subjects and parents able to commit to the intensive therapy program for a period of 3 weeks

Exclusion Criteria:

* Children who had sustained previous orthopedic surgery or botulinum toxin A injection in the UL within 6 months prior to study entry were excluded.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Changes in the Assisting Hand Assessment | Baseline (T0, 1week before beginning of Study) ;T1 (within 1 week after the end of the training/control period); T1 plus (within 1 week after the end of training for waitlist group), T2 and T3 (8weeks after T1 or T1/plus) T3 (16 weeks after T2)
  This assessment measures upper limb function during bimanual activities. The test evaluates spontaneous use of assisting hand during a semi-structured session with specific toys or tasks with objects requiring bimanual handling

SECONDARY OUTCOMES:
Changes in Box and Block Test | Baseline (T0, 1week before beginning of Study) ;T1 (within 1 week after the end of the training/control period); T1 plus (within 1 week after the end of training for waitlist group), T2 and T3 (8weeks after T1 or T1/plus) T3 (16 weeks after T2)
  : it measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations from childhood to adults.
Changes in Melbourne Assessment of Unilateral Upper Limb Function | Baseline (T0, 1week before beginning of Study) ;T1 (within 1 week after the end of the training/control period); T1 plus (within 1 week after the end of training for waitlist group), T2 and T3 (8weeks after T1 or T1/plus) T3 (16 weeks after T2)
  It is criterion-referenced test that measures unilateral upper extremity quality of movement in subjects with neurological impairments
Changes in ABILHAND-kids | Baseline (T0, 1week before beginning of Study) ;T1 (within 1 week after the end of the training/control period); T1 plus (within 1 week after the end of training for waitlist group), T2 and T3 (8weeks after T1 or T1/plus) T3 (16 weeks after T2)
  a semi-structured item-response questionnaire that measures manual ability according to an caregiver's perceived difficulty performing daily bimanual tasks.

OTHER OUTCOMES:
Participation and Environment Measure - Children and Youth (PEM-CY) | Baseline (T0) and T3 (16 weeks after T2)
  it is a measure that evaluates participation in the home, at school, and in the community, alongside environmental factors within each of these settings.
Cerebral Palsy Quality of Life Questionnaire | Baseline (T0) and T3 (16 weeks after T2)
  These instruments are useful for evaluating interventions designed to improve the lives of children and adolescents
Quantitative measurement of reaching and grasping capabilities by means of a sensorized object that allow different grasping tasks | Baseline (T0, 1week before beginning of Study) ;T1 (within 1 week after the end of the training/control period); T1 plus (within 1 week after the end of training for waitlist group), T2 and T3 (8weeks after T1 or T1/plus) T3 (16 weeks after T2)
  The sensorized object allows to perform three different tasks at increasing level of difficulties (unimanual lifting, bimanual placing near and bimanual cooperation, holding and pulling)
Quantitative Changes in upper limbs activities detected with Actigraph GXT3+ during AHA | Baseline (T0, 1week before beginning of Study); T1 (within 1 week after the end of the training/control period); T1 plus (within 1 week after the end of training for waitlist group), T2 and T3 (8weeks after T1 or T1/plus) T3 (16 weeks after T2)
  Actigraph GXT3+ worn during AHA assessments
Changes in daily life activities detected with Actigraph GXT3+ | During training and/or standard period (from T0 to T1 and/or T1 to T1plus) (T0,1week before beginning of Study); T1 (within 1 week after the end of the training/control period); T1 plus (within 1 week after the end of training for waitlist group)
  Quantitative measurement of daily manual activities

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Stella Maris Foundation, Calambrone, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sgandurra G, Ferrari A, Cossu G, Guzzetta A, Biagi L, Tosetti M, Fogassi L, Cioni G. Upper limb children action-observation training (UP-CAT): a randomised controlled trial in hemiplegic cerebral palsy. BMC Neurol. 2011 Jun 28;11:80. doi: 10.1186/1471-2377-11-80. PMID 21711525
- [Background] Sgandurra G, Ferrari A, Cossu G, Guzzetta A, Fogassi L, Cioni G. Randomized trial of observation and execution of upper extremity actions versus action alone in children with unilateral cerebral palsy. Neurorehabil Neural Repair. 2013 Nov-Dec;27(9):808-15. doi: 10.1177/1545968313497101. Epub 2013 Jul 25. PMID 23886886
- [Derived] Beani E, Menici V, Ferrari A, Cioni G, Sgandurra G. Feasibility of a Home-Based Action Observation Training for Children With Unilateral Cerebral Palsy: An Explorative Study. Front Neurol. 2020 Feb 28;11:16. doi: 10.3389/fneur.2020.00016. eCollection 2020. PMID 32180754
- [Derived] Sgandurra G, Cecchi F, Beani E, Mannari I, Maselli M, Falotico FP, Inguaggiato E, Perazza S, Sicola E, Feys H, Klingels K, Ferrari A, Dario P, Boyd RN, Cioni G. Tele-UPCAT: study protocol of a randomised controlled trial of a home-based Tele-monitored UPper limb Children Action observation Training for participants with unilateral cerebral palsy. BMJ Open. 2018 May 14;8(5):e017819. doi: 10.1136/bmjopen-2017-017819. PMID 29764869